CLINICAL TRIAL: NCT03744182
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of HM15211(Efocipegtrutide) in Obese Subjects With NAFLD
Brief Title: A Study of Multiple Doses of HM15211(Efocipegtrutide) in Obese Subjects With NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HM-TRIA-102
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15211 (Experimental)
  Interventions: Drug: HM15211
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of HM15211

INTERVENTIONS:
Drug: HM15211 — A sterile solution of HM15211 contained in pre-filled syringes
  Arms: HM15211
Drug: Placebo of HM15211 — A sterile, matching solution in pre-filled syringes
  Arms: Placebo

SUMMARY:
This study is a phase 1 study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of HM15211 in obese subjects with NAFLD

DETAILED DESCRIPTION:
This study will be single-blind and conducted in up to 6 cohorts comprising a total of up to 72 obese subjects with NAFLD. Each cohort will enroll subjects to ensure that at least 12 subjects per cohort will complete the study. Subjects will be randomized to investigational product (IP) or placebo in a 3:1 ratio via an Interactive Web Response System (IWRS). Per cohort (n=12 subjects), 9 subjects will be randomized to IP and 3 subjects to placebo. Cohorts may partially overlap after at least 9 subjects have completed 2-4 weeks of treatment (2 weeks of treatment is reached at Visit week 3) and a dose escalation decision has been made. Study drug will be administered weekly over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 30 kg/m2
* Waist circumference ≤ 57 inches
* Fasting Plasma Glucose < 7 mmol/L (126 mg/dL)
* HbA1c < 6.5%
* Controlled Attenuation Parameter ≥ 300 dB/m by FibroScan
* Liver fat by MRI-PDFF ≥ 10%.

Exclusion Criteria:

* A history of or active chronic liver disease due to alcohol, auto-immune, HIV, HBV or active HCV-infection or NASH disease
* Any history of clinically significant chronic liver disease including esophageal varices, ascites, encephalopathy or any hospitalization for treatment of chronic liver disease; or Model for End Stage Liver Disease (MELD) ≥ 10
* Previous surgical treatment for obesity
* Uncontrolled hypertension
* Any weight control treatment
* History or current diagnosis of acute or chronic pancreatitis or factors for pancreatitis
* History of major depression, anxiety, suicidal behavior or attempts, or other psychiatric disorder requiring medical treatment
* History or current diagnosis of heart disease
* Presence of clinically significant ECG findings
* History of renal disease or abnormal kidney function tests
* History of alcohol or illicit drug abuse
* Daily heavy use of cigarettes or any tobacco product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento Inc., Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment was November 1st, 2018. Last subject was enrolled on March 3rd, 2020.
Groups:
- 0.01 mg/kg HM15211: HM15211: A sterile solution of HM15211 contained in pre-filled syringes
  0.01 mg/kg HM15211
- 0.02 mg/kg HM15211: HM15211: A sterile solution of HM15211 contained in pre-filled syringes 0.02 mg/kg HM15211
- 0.04 mg/kg HM15211: HM15211: A sterile solution of HM15211 contained in pre-filled syringes 0.04 mg/kg HM15211
- 0.06 mg/kg HM15211: HM15211: A sterile solution of HM15211 contained in pre-filled syringes 0.06 mg/kg HM15211
- 0.08 mg/kg HM15211: HM15211: A sterile solution of HM15211 contained in pre-filled syringes 0.08 mg/kg HM15211
Period: Overall Study
Arm/Group | 0.01 mg/kg HM15211 | 0.02 mg/kg HM15211 | 0.04 mg/kg HM15211 | 0.06 mg/kg HM15211 | 0.08 mg/kg HM15211 | Placebo
Started | 9 | 10 | 12 | 9 | 9 | 17
Completed | 9 | 10 | 10 | 9 | 8 | 15
Not Completed | 0 | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- HM15211 0.01 mg/kg; HM15211 0.02 mg/kg; HM15211 0.04 mg/kg; HM15211 0.06 mg/kg; HM15211 0.08 mg/kg: HM15211: A sterile solution of HM15211 contained in pre-filled syringes
- Total: Total of all reporting groups
Arm/Group | HM15211 0.01 mg/kg | HM15211 0.02 mg/kg | HM15211 0.04 mg/kg | HM15211 0.06 mg/kg | HM15211 0.08 mg/kg | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 12 | 9 | 9 | 17 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 8 | 3 | 3 | 9 | 33
  Male | 6 | 3 | 4 | 6 | 6 | 8 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Hispanic or Latino | 7 | 10 | 11 | 8 | 7 | 14 | 57
  Ethnicity : Not Hispanic or Latino | 2 | 0 | 1 | 1 | 2 | 3 | 9
  Race : White | 8 | 10 | 10 | 9 | 6 | 15 | 58
  Race : Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Race : Black or African American | 0 | 0 | 1 | 0 | 2 | 2 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race: Multiple | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 12 | 9 | 9 | 17 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Cardiovascular events, rash/inflammatory dermatitis and other skin disorders, GI events, and gallstone formation [cholelithiasis] were managed following a separate AE guidance document
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HM15211 0.01 mg/kg | HM15211 0.02 mg/kg | HM15211 0.04 mg/kg | HM15211 0.06 mg/kg | HM15211 0.08 mg/kg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17
Participants | 7 | 9 | 9 | 8 | 6 | 8

2. Primary Outcome: Incidence of Clinical Renal Function Lab Abnormalities
Description: Observed Values and Change from Baseline in Renal Function of Urea Nitrogen
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HM15211 0.01 mg/kg | HM15211 0.02 mg/kg | HM15211 0.04 mg/kg | HM15211 0.06 mg/kg | HM15211 0.08 mg/kg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17
mmol/L | -1.111 (0.7240) | -0.238 (0.7142) | 0.036 (1.1350) | -0.754 (0.7242) | -0.893 (0.5414) | 0.190 (1.4962)

3. Primary Outcome: Vital Signs
Description: Change from baseline in vital signs (Systolic Blood)
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HM15211 0.01 mg/kg | HM15211 0.02 mg/kg | HM15211 0.04 mg/kg | HM15211 0.06 mg/kg | HM15211 0.08 mg/kg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17
mmHg | 7.2 (14.96) | 7.1 (12.64) | -0.7 (13.33) | -3.3 (8.67) | -4.5 (18.80) | 2.2 (12.27)

4. Primary Outcome: 12-lead ECG
Description: Change from baseline in 12-lead ECG; the primary ECG endpoint was QTcF
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | HM15211 0.01 mg/kg | HM15211 0.02 mg/kg | HM15211 0.04 mg/kg | HM15211 0.06 mg/kg | HM15211 0.08 mg/kg | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17
milliseconds | 4.2 (7.79) | 1.3 (9.51) | -1.3 (7.14) | 0 (3.59) | -2.2 (9.02) | 2.5 (4.83)

5. Secondary Outcome: Body Mass Index
Description: Change of Body Mass Index from baseline to 12 weeks after IP injection
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | 0.01 mg/kg HM15211 | 0.02 mg/kg HM15211 | 0.04 mg/kg HM15211 | 0.06 mg/kg HM15211 | 0.08 mg/kg HM15211 | Placebo
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 9 | 17
kg/m2 | 35.46 (3.835) | 32.91 (2.936) | 37.86 (6.254) | 40.13 (7.113) | 35.74 (3.796) | 34.61 (3.521)

ADVERSE EVENTS:
Time Frame: 23 weeks
Description: All AEs were collected over 23 weeks in safety analysis set.
Arm/Group | 0.01 mg/kg HM15211 | 0.02 mg/kg HM15211 | 0.04 mg/kg HM15211 | 0.06 mg/kg HM15211 | 0.08 mg/kg HM15211 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/12 | 0/9 | 0/9 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/12 | 0/9 | 0/9 | 0/17
Other Adverse Events (participants affected / at risk) | 7/9 | 9/10 | 9/12 | 8/9 | 6/9 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.01 mg/kg HM15211 (N=9) | 0.02 mg/kg HM15211 (N=10) | 0.04 mg/kg HM15211 (N=12) | 0.06 mg/kg HM15211 (N=9) | 0.08 mg/kg HM15211 (N=9) | Placebo (N=17)
nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 2 | 0 | 0 | 3
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 1 | 2 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03744182/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT03744182/SAP_001.pdf